CLINICAL TRIAL: NCT01125553
Title: A Trial to Test for Bioequivalence Between Two NN5401 Formulations in Healthy Subjects
Brief Title: A Comparison Between Two Formulations of NN5401 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN5401-1980; U1111-1113-7011 (Other: WHO)
Record Dates: First submitted 2010-05-07; First posted 2010-05-18 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp B (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- IDegAsp F (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Each subject will be allocated to two single injections of trial product on two separate dosing visits with each of the two insulin degludec/insulin aspart formulations. The trial products will be administered as a subcutaneous injection (under the skin).

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of the trial is to compare the exposure of two formulations of insulin degludec/insulin aspart (NN5401) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Considered generally healthy upon completion of medical history, physical examination, vital signs and electrocardiogram (ECG), as judged by the physician
* Body mass index between 18.0 and 27.0 kg/m^2 (both inclusive)

Exclusion Criteria:

* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to trial start
* Smoker (defined as a subject who is smoking more than 5 cigarettes or the equivalent per day)
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Area under the serum insulin degludec concentration-time curve | from 0 to 120 hours after single-dose
Maximum observed serum insulin degludec concentration | from 0 to 120 hours after single-dose
Area under the serum insulin aspart concentration-time curve | from 0 to 12 hours after single-dose
Maximum observed serum insulin aspart concentration | from 0 to 12 hours after single-dose

SECONDARY OUTCOMES:
Time to maximum observed serum insulin degludec concentration | from 0 to 120 hours after single-dose
Time to maximum observed serum insulin aspart concentration | from 0 to 12 hours after single-dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Clinical Trial Call Center, Chula Vista, California, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com